CLINICAL TRIAL: NCT00669682
Title: T-wave Alternans and Intrathoracic Impedance Measurements
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jose M. Dizon, Assoc Professor of Clinical, Department of Cardiology, Columbia University
Other Study IDs: AAAC5529
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Congestive Heart Failure; Arrhythmias
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: The study group will include Class III to IV heart failure patients followed in the device clinic that have a chronically implanted (more than 90 days) Medtronic biventricular defibrillator with the ability to monitor intrathoracic impedance.
  Interventions: Other: Congestive heart failure

INTERVENTIONS:
Other: Congestive heart failure — Spontaneous occurrence of fluid overload.

SUMMARY:
T-wave alternans is a test that is currently being used to risk stratify patients with structural heart disease for sudden cardiac death. The mechanism of T-wave alternans is unclear, but may share a common abnormality with conditions of cardiac fluid overload such as heart failure, which is altered intracellular calcium handling. Current Medtronic implantable defibrillators have the capability of monitoring cardiac fluid status via transthoracic impedance measurements.

The purpose of this study is to determine if a correlation exists between T-wave alternans status and cardiac volume status, as determined by transthoracic impedance measurements. Secondarily, the study seeks to examine the relationship between arrhythmia frequency and T-wave alternans or cardiac volume status.

ELIGIBILITY:
Inclusion Criteria:

* Class III or IV heart failure patients with a chronically implanted Medtronic biventricular defibrillator system capable of monitoring intrathoracic fluid volume.

Exclusion Criteria:

* no active ischemia or pulmonary edema, atrial fibrillation, complete heart block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Class III or IV heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Dizon, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 patients enrolled from device clinic between 8/14/08 and 2/11/11
Period: Overall Study
Arm/Group | Group A
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group A
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Positive Twave Studies and Concurrent Positive Optivol Measurement
Description: We wanted to examine whether positive Optivol status corresponded to a higher likelihood of a positive T wave study. The T wave alternans result is determined by a proprietary device that measures T wave and reports the result as negative, positive, or indeterminate. The Optivol measurement is obtained through transthoracic impedance values in the implanted device. We investigated the correlation between Optivol status and T wave alternans status.
Time Frame: upto 3 years
Measure: Number; unit: participants
Groups:
- Positive Optivol Status: These patients have transthoracic impedance measurements that suggest fluid overload
- Negative Optivol Status: These patients have transthoracic impedance measurements that do not suggest fluid overload
Arm/Group | Positive Optivol Status | Negative Optivol Status
Number analyzed (Participants) | 3 | 6
participants
  Positive T wave alternans | 1 | 1
  Negative T wave alternans | 2 | 5

ADVERSE EVENTS:
Arm/Group | Group A
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No